CLINICAL TRIAL: NCT01945905
Title: Cost-effectiveness of Two Forms of Delivery of Directly Observed Treatment in a Demonstration Area of the DOTS Strategy in Colombia
Brief Title: Cost-effectiveness of Two Forms of DOTS in a Demonstration Area of the DOTS Strategy in Colombia
Acronym: DOTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FES (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Sandra Lorena Girón Vargas, Msc Epidemiologist, Fundación FES
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FES02013
Record Dates: First submitted 2013-09-09; First posted 2013-09-19 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis; Adherence, medication; Patient compliance
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Medication Adherence; Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extramural (Experimental): Extramural medication delivery and supervision
  Interventions: Other: Extramural
- Intramural (Active Comparator): Intramural medication delivery and supervision
  Interventions: Other: Intramural

INTERVENTIONS:
Other: Intramural — Under this alternative, the patients will receive treatment with direct observation from health team. Treatment will be provided for free
  Arms: Intramural
Other: Extramural — In this form the medication will be given by a health worker in the place chosen by patients. This option will be delivered to patients with newly diagnosed pulmonary TB without hospitalization criteria
  Arms: Extramural

SUMMARY:
* Tuberculosis ( TB ) remains a major global public health problems and actions to ensure the diagnosis and complete treatment of all cases is the priority for the control of this disease. Despite the availability of effective anti-tuberculosis medications, there are still high levels of nonadherence to treatment. The nonadherence increases the morbidity and mortality of patients, decreases the cure rate, increases the community transmission and the increase of chronically ill patients enables the emergence of multi - drug resistant and increases treatment costs.
* Despite the knowledge about different forms of cost-effective delivery of DOT (directly observed treatment), recognition of the need to establish the DOT strategy related to the context from local studies, in Colombia and in Cali we hadn't had made studies similar than this one that establish the cost and results of the current DOT delivery strategy and to identify other ways to improve adherence and cure rate for the TB patients at reasonable cost for both: health services and families
* Therefore, this research aims to compare the cost -effectiveness of current DOT delivery method with an alternative extra- institutional delivery of anti -TB treatment in urban areas of Cali. A cost-effectiveness study was conducted from the institutional and familiar perspective with prospective information collection.

DETAILED DESCRIPTION:
We compared two strategies for anti- TB treatment delivery: one institutional in which patients went to health institutions to receive treatment and other extra- institutional in which the medication was delivered in the place of choice for treating patients.

Measuring the effectiveness ( compliance and cure ) was made from a controlled clinical trial , randomized , partially blinded . The measurement of family and institutional costs , direct and indirect , will be based on the activities.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (non-pregnant)
* 15 years of age and older
* Living in urban area (Cali)
* New diagnosed patients (TB)
* In conditions to give survey information
* Patients without hemoptysis and special conditions like: hepatic disease, renal failure, diabetes, hypertension, HIV/AIDS and negative test for pulmonary tuberculosis

Exclusion Criteria:

* Not written informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2009-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Compliance with treatment | Participants will be followed for the duration of the treatment, an expected average of six months
  Total of patients who completed de treatment

SECONDARY OUTCOMES:
Cured patients | Participants will be followed for the duration of the treatment, an expected average of six months
  Total number of patients who completed the treatment and had the last or the two last smear negative and had negative cultures at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Giron, Msc Epi, Principal Investigator — Fundación FES; Julio C Mateus, Msc Epi, Principal Investigator — Fundación FES
Locations (1):
- Secretaria de Salud Publica Municipal de Cali, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Moulding T, Mateus-Solarte JC, Carvajal-Barona R. Factors predictive of adherence to tuberculosis treatment, Valle del Cauca, Colombia. Int J Tuberc Lung Dis. 2009 Mar;13(3):416-7; author reply 417-8. No abstract available. PMID 19275807
- [Background] Pablos-Mendez A, Knirsch CA, Barr RG, Lerner BH, Frieden TR. Nonadherence in tuberculosis treatment: predictors and consequences in New York City. Am J Med. 1997 Feb;102(2):164-70. doi: 10.1016/s0002-9343(96)00402-0. PMID 9217566
- [Background] Burman WJ, Cohn DL, Rietmeijer CA, Judson FN, Sbarbaro JA, Reves RR. Noncompliance with directly observed therapy for tuberculosis. Epidemiology and effect on the outcome of treatment. Chest. 1997 May;111(5):1168-73. doi: 10.1378/chest.111.5.1168. PMID 9149565
- [Background] O'Boyle SJ, Power JJ, Ibrahim MY, Watson JP. Factors affecting patient compliance with anti-tuberculosis chemotherapy using the directly observed treatment, short-course strategy (DOTS). Int J Tuberc Lung Dis. 2002 Apr;6(4):307-12. PMID 11936739
- [Background] Jaiswal A, Singh V, Ogden JA, Porter JD, Sharma PP, Sarin R, Arora VK, Jain RC. Adherence to tuberculosis treatment: lessons from the urban setting of Delhi, India. Trop Med Int Health. 2003 Jul;8(7):625-33. doi: 10.1046/j.1365-3156.2003.01061.x. PMID 12828545
- [Background] Clarke M, Dick J, Bogg L. Cost-effectiveness analysis of an alternative tuberculosis management strategy for permanent farm dwellers in South Africa amidst health service contraction. Scand J Public Health. 2006;34(1):83-91. doi: 10.1080/14034940510032220. PMID 16449048
- [Background] Islam MA, Wakai S, Ishikawa N, Chowdhury AM, Vaughan JP. Cost-effectiveness of community health workers in tuberculosis control in Bangladesh. Bull World Health Organ. 2002;80(6):445-50. PMID 12132000
- [Background] Sinanovic E, Floyd K, Dudley L, Azevedo V, Grant R, Maher D. Cost and cost-effectiveness of community-based care for tuberculosis in Cape Town, South Africa. Int J Tuberc Lung Dis. 2003 Sep;7(9 Suppl 1):S56-62. PMID 12971655
- [Background] Lwilla F, Schellenberg D, Masanja H, Acosta C, Galindo C, Aponte J, Egwaga S, Njako B, Ascaso C, Tanner M, Alonso P. Evaluation of efficacy of community-based vs. institutional-based direct observed short-course treatment for the control of tuberculosis in Kilombero district, Tanzania. Trop Med Int Health. 2003 Mar;8(3):204-10. doi: 10.1046/j.1365-3156.2003.00999.x. PMID 12631309
- [Background] Khan MA, Walley JD, Witter SN, Imran A, Safdar N. Costs and cost-effectiveness of different DOT strategies for the treatment of tuberculosis in Pakistan. Directly Observed Treatment. Health Policy Plan. 2002 Jun;17(2):178-86. doi: 10.1093/heapol/17.2.178. PMID 12000778
- [Background] Okello D, Floyd K, Adatu F, Odeke R, Gargioni G. Cost and cost-effectiveness of community-based care for tuberculosis patients in rural Uganda. Int J Tuberc Lung Dis. 2003 Sep;7(9 Suppl 1):S72-9. PMID 12971657
- [Background] Wandwalo E, Robberstad B, Morkve O. Cost and cost-effectiveness of community based and health facility based directly observed treatment of tuberculosis in Dar es Salaam, Tanzania. Cost Eff Resour Alloc. 2005 Jul 14;3:6. doi: 10.1186/1478-7547-3-6. PMID 16018806
- [Background] Elamin EI, Ibrahim MI, Sulaiman SA, Muttalif AR. Cost of illness of tuberculosis in Penang, Malaysia. Pharm World Sci. 2008 Jun;30(3):281-6. doi: 10.1007/s11096-007-9185-0. Epub 2008 Jan 18. PMID 18204974